CLINICAL TRIAL: NCT05477693
Title: A Randomized, Double-blind, Positive-controlled Phase Ⅳ Clinical Trial to Evaluate the Immunogenicity and Safety of 23-valent Pneumococcal Polysaccharide Vaccine in Population Aged 2 Years and Older
Brief Title: Immunogenicity and Safety of 23-valent Pneumococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO-PPV-4002
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-04

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 1200 participants(including 600 subjects aged 2~17 years,240 subjects aged 18~59 years and 360 subjects aged 60 years and above)received one dose of 23-valent pneumococcal polysaccharide vaccine manufactured by Sinovac Biotech Co., Ltd
  Interventions: Biological: Experimental 23-valent PPV
- Control Group (Active Comparator): 600 participants(including 300 subjects aged 2~17 years,120 subjects aged 18~59 years and 180 subjects aged 60 years and above)received one dose of 23-valent pneumococcal polysaccharide vaccine manufactured by Merck Sharp & Dohme.
  Interventions: Biological: Control 23-valent PPV

INTERVENTIONS:
Biological: Experimental 23-valent PPV — The investigational vaccine was manufactured by Sinovac Biotech Co., Ltd.25μg each for serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B,17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in 0.5 mL of sodium chloride, sodium dihydrogen phosphate and disodium hydrogen phosphate per injection.
  Arms: Experimental Group
Biological: Control 23-valent PPV — The control vaccine was manufactured by Merck Sharp & Dohme, Ltd. Purified capsular polysaccharides from 23 Streptococcus in 0.5 mL of pneumoniae types 0.25% phenol and sodium chloride.
  Arms: Control Group

SUMMARY:
This is a randomized, double-blind, positive-controlled phase Ⅳ clinical trial of 23-valent pneumococcal polysaccharide vaccine manufactured by Sinovac Biotech Co., Ltd.The purpose of this study is to evaluate the immunogenicity and safety of 23-valent pneumococcal polysaccharide vaccine in population aged 2 years and older.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, positive-controlled phase Ⅳ clinical trial to evaluate the immunogenicity and safety of 23-valent pneumococcal polysaccharide vaccine in population aged 2 years and older.The experimental vaccine was manufactured by Sinovac Biotech Co., Ltd,the control vaccine was manufactured by Merck Sharp & Dohme.A total of 1800 subjects including 900 subjects aged 2~17 years,360 subjects aged 18~59 years and 540 subjects aged 60 years and above will be enrolled.Subjects in each age group will be randomly divided into two groups according to the ratio of 2:1, and received one dose of experimental vaccine or control vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 years and above in stable health;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 8-17 years, both subjects and guardians need to sign the informed consent form.If the subject aged 16 to 17 years with full capacity for civil conduct and his/her labor income is his/her main source of living, the informed consent can be signed only by the subject himself/herself);
* Proven legal identity.

Exclusion Criteria:

* Have received any pneumococcal vaccine;
* History bacterial pneumonia or invasive pneumococcal infectious diseases caused by pneumococci and confirmed by culture.
* Women of childbearing age (menarche to premenopause) are pregnant (including positive urine pregnancy test), breastfeeding or planning pregnancy within 1 month;
* History of asthma, allergy to vaccines or vaccine components, and serious adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema;
* Severe chronic diseases,such as severe cardiovascular diseases, hypertension(Systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg) and diabetes that cannot be controlled by drugs, liver or kidney diseases,malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* A long history of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs within 30 days prior to receiving the investigational vaccine;
* Receipt of attenuated live vaccines or COVID-19 vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 3 days prior to the study;
* Underarm body temperature before vaccination>37.0°C;
* The subjects participated in other clinical trials during the follow-up period or will be planned to participate other clinical trials within 1 months;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-Seroconversion rate (2-fold increase rate) | 30 days after vaccination
  Seroconversion rate (2-fold increase rate)for serotype specificity (3, 6B, 14, 19A, 19F, 23F) of pneumococcal immunoglobulin G (IgG) antibody 30 days after vaccination.

SECONDARY OUTCOMES:
Immunogenicity index-Geometric Mean Concentration (GMC) | 30 days after vaccination
  Geometric Mean Concentration (GMC) for serotype specificity (3, 6B, 14, 19A, 19F, 23F) of pneumococcal IgG antibody 30 days after vaccination.
Immunogenicity index-Geometric Mean Increase (GMI) | 30 days after vaccination
  Geometric Mean Increase (GMI) for serotype specificity (3, 6B, 14, 19A, 19F, 23F) of pneumococcal IgG antibody 30 days after vaccination.
Immunogenicity index-Seroconversion rate | 30 days after vaccination
  Seroconversion rate for serotype specificity （1、2、4、5、7F、8、9N、9V、10A、11A、12F、15B、17F、18C、20、22F and 33F）of pneumococcal IgG antibody 30 days after vaccination.
Immunogenicity index-GMC | 30 days after vaccination
  Geometric Mean Concentration (GMC) for serotype specificity （1、2、4、5、7F、8、9N、9V、10A、11A、12F、15B、17F、18C、20、22F and 33F）of pneumococcal IgG antibody 30 days after vaccination.
Immunogenicity index-GMI | 30 days after vaccination
  Geometric Mean Increase (GMI) for serotype specificity （1、2、4、5、7F、8、9N、9V、10A、11A、12F、15B、17F、18C、20、22F and 33F）of pneumococcal IgG antibody 30 days after vaccination.
Safety index-Incidence of adverse reactions | Within 30 days after vaccination
  Incidence of adverse reactions within 30 days after vaccination.
Safety index-incidence of adverse reactions | Within 7 days after vaccination
  Incidence of adverse reactions within 7 days after vaccination
Safety index-Incidence of serious adverse events | Within 30 days after vaccination
  Incidence of serious adverse events within 30 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Hu, Principal Investigator — Shanxi Provincial Center for Disease Prevention and Control
Locations (1):
- Linwei District Center for Disease Control and Prevention, Weinan, Shanxi, China